CLINICAL TRIAL: NCT07142564
Title: Carrier Care: An Innovative Approach to Support Small Babies in the NICU
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Lisa Grisham, PhD, DNP, NNP-BC, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006871
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Group 1: Carrier Care (CC) Followed by Skin-to-Skin Care (SSC) Followed by Family Choice; Group 2: Skin-to-Skin Care (SSC) Followed by Carrier Care (CC) Followed by Family Choice
Keywords: carrier care; skin-to-skin care (ssc); infant carrier; babywearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1: Carrier Care (CC) followed by Skin-to-Skin Care (SSC) followed by Family Choice (Other): Carrier Care
  Interventions: Other: Carrier Care (CC)

INTERVENTIONS:
Other: Carrier Care (CC) — Carrier care uses an infant carrier to secure the infant to the caregiver, while SSC does not have a securing device. The caregiver holds the infant with their arms.

SUMMARY:
The significance of skin-to-skin care (SSC) for neonatal infants is well-documented, highlighting its benefits for both the infant and the caregiver. The World Health Organization (WHO) has emphasized the necessity of positioning the infant on the mother after birth in a manner to prevent Sudden Unexpected Postnatal Collapse (SUPC) and accidental drops and falls. SSC is also recommended for 8 hours a day for the first few weeks of life to promote a secure attachment in the infant and bonding with the caregiver.

Despite these established benefits, some families hesitate to engage in skin-to-skin care (SSC) because it is often only done in private settings and requires the caregiver to use their arms to hold the infant in place. Babywearing, or holding the infant to the body of the caregiver using a cloth or infant carrying device, can promote prolonged contact between the caregiver and infant without requiring the caregiver to hold the infant in place with their arms. Babywearing can also be done in more public settings (e.g., grocery store) as the caregiver can remain clothed during babywearing. The purpose of this study is to investigate whether babywearing using a babywearing device, referred to in this study as Carrier Care (CC), is at least as feasible and effective as SSC. This research will evaluate several physiological parameters of the infant, including cardiorespiratory stability, thermoregulation, and oxygen saturation levels. Certified babywearing educators will instruct research participants to ensure proper use of baby carriers and the safety of infants as outlined by the current hospital policy for babywearing.

This study will utilize an amplitude-integrated electroencephalogram (aEEG), a non-invasive, bedside monitoring tool commonly used in neonatal intensive care units (NICUs) to assess brain activity, particularly in premature infants. The aEEG provides a simplified and continuous recording of cortical activity, offering valuable insights into neurological development, including sleep-wake cycling. In this study, the aEEG will be used to evaluate the presence of sleep-wake patterns as a proxy for brain maturation. Data will be collected by placing EEG electrodes on the infant for a total duration of 12 hours: 4 hours prior to the intervention (baseline), 4 hours during the intervention (defined as skin-to-skin contact or carrier care), and 4 hours post-intervention. Recordings will occur on day 3 of the randomized activity to assess potential changes in brain activity associated with the intervention during this critical period of neurodevelopment. Dau 4 or 5 will be used as backup.

DETAILED DESCRIPTION:
A large body of research on skin-to-skin contact (SSC), particularly for preterm infants, provides robust evidence that it benefits both mothers and infants (Koreti & Muntode Gharde, 2022). Premature infants in the NICU are often separated from their caregivers and placed into an otherwise artificial environment, leading to neurological, sociological, and psychological consequences, along with the impacts of being born prematurely. In addition to positive outcomes, it is notable that SSC is a safe intervention. For example, one review found no negative impact on vital signs or any reports of adverse events before, during, or after SSC (Bisanalli et al., 2023). Overall, SSC shortens hospital stays in the NICU, lowers risks for neonatal infection, increases weight gain, lowers cortisol levels, increases feeding tolerance, and helps with thermoregulation and homeostasis while being safe for the infants and their caregivers participating (Azevedo et al., 2012; Cristóbal Cañadas et al., 2022).

Research on babywearing (close physical contact while clothed or extended arms-free holding) is growing, but a recent scoping review indicates positive biological and behavioral effects for both mothers and infants (Grisham et al., 2023). This research team has previously demonstrated that babywearing effectively increases infant and caregiver comfort among infants diagnosed with Neonatal Abstinence Syndrome (Williams et al., 2020). We recently replicated this finding (Rankin et al., 2024), and also found that babywearing was perceived by nurses as helpful in the care and treatment of these infants (Williams et al., 2021). From the caregiver's perspective, babywearing helps with the tasks of parenting (e.g., calming the infant, putting the infant to sleep), increases bonding time, and is convenient (i.e., provides hands-free to complete other tasks) (Williams, 2020). Our research question is guided by the perspective that if babywearing can closely approximate the benefits of SSC, it would provide a more comfortable and convenient alternative to SSC and potentially extend the benefits by allowing for a greater amount of time spent in close physical proximity.

This project investigates the application of amplitude-integrated electro-encephalography (aEEG) to monitor brain activity and sleep-wake cycling in premature and term neonates in NICU settings. Continuous EEG monitoring for at least 2-3 hours is essential to capture both wakefulness and all stages of sleep. It typically utilizes a compressed display to evaluate slow activity and asynchronies critical in neonatal recordings (Mizrahi & Kellaway, 2017). The aEEG provides a simplified, bedside tool for long-term monitoring of cerebral function, allowing detection of seizures and assessment of background brain activity patterns (Hellström-Westas et al., 2006) (Shellhaas et al., 2023). aEEG has proven especially useful in neonates with seizures, offering early prediction of neurodevelopmental outcomes based on patterns observed within the first 24 hours after birth (Shellhaas et al., 2023). The early presence of sleep-wake cyclicity on aEEG strongly predicts favorable brain imaging outcomes, while delayed or absent cyclicity is associated with severe abnormalities (Bruns et al., 2017).

Preterm infants show altered sleep patterns compared to term infants, with shorter sleep cycles and increased REM sleep, both of which are essential for brain maturation (Bandyopadhyay et al., 2017). Disrupted or insufficient sleep in NICU infants has been linked to short-term physiological alterations and long-term developmental delays, reinforcing the importance of protecting and promoting sleep quality (Gale et al., 2012; Gertner et al., 2012). aEEG is safe, well-tolerated even by extremely preterm infants, and can be interpreted by neonatal staff due to its simplicity and strong interrater reliability (Hellström-Westas et al., 2006; Toet et al., 2006). This research supports the advancement of non-invasive, accessible neuro-monitoring to guide care and improve neurodevelopmental outcomes in high-risk neonatal populations.

Inclusion Criteria for Infants

Participants for this study will include neonates:

* admitted to the hospital
* who have an estimated length of stay equal to or greater than fifteen (15) days
* weighing greater than or equal to 1800 grams at the time of enrollment
* that are medically stable (free of significant apnea, bradycardia, or desaturations) within the past 48 hours

Inclusion Criteria for Caregivers

Caregivers of infant participants for this study will include:

* caregivers must be 18 years or older,
* those willing to comply with the study protocol, specifically to participate daily in carrier care (CC) and skin-to-skin care (SSC) for fifteen (15) consecutive days.

Exclusion Criteria for Infants and Caregivers

Study participants who will be excluded from this study include:

* infants who require oxygen therapy or positive pressure respiratory support
* infants who have central intravenous lines (e.g., Broviac or peripherally inserted central catheter)
* caregivers who are prisoners
* caregivers who cannot read or speak English

ELIGIBILITY:
Inclusion Criteria:

Neonates who:

* are admitted to the hospital
* who have an estimated length of stay equal to or greater than fifteen (15) days
* weighing greater than or equal to 1800 grams at the time of enrollment
* that are medically stable (free of significant apnea, bradycardia, or desaturations) within the past 48 hours

Exclusion Criteria:

* infants who require oxygen therapy or positive pressure respiratory support
* infants who have central intravenous lines (e.g., Broviac or peripherally inserted central catheter)
* caregivers who are prisoners
* caregivers who cannot read or speak English

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Stability | From enrollment to study completion at 15 days.
  Evaluate the cardiorespiratory stability of the infant during carrier care (CC) or skin-to-skin care (SSC).

SECONDARY OUTCOMES:
Thermoregulation | From enrollment to study completion at 15 days.
  Evaluate the thermal stability of the infant before and after carrier care (CC) and skin-to-skin care (SSC) as measured by an axillary temperature reading of 36.5-37.5°C.

IPD SHARING:
Plan to Share IPD: Undecided
Still developing the plan